CLINICAL TRIAL: NCT04370444
Title: Pathways for Patient-centered Diagnosis and Management of Endometriosis-associated Deep Dyspareunia: A Pilot Randomized Trial
Brief Title: Pathways for Patient-centered Diagnosis and Management of Endometriosis-associated Deep Dyspareunia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BC Women's Hospital & Health Centre (Other)
Responsible Party: Principal Investigator, Paul Yong, Principal Investigator, BC Women's Hospital & Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H19-00294
Record Dates: First submitted 2020-04-23; First posted 2020-05-01 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis-related Pain; Dyspareunia Deep
Keywords: endometriosis; dyspareunia; sexual distress; buffer
MeSH Terms: conditions — Endometriosis; Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (PLR) (Experimental): Participants will be given the OhNut Phallus Length Reducer (PLR) for use during the study period.
  Interventions: Device: Phallus Length Reducer; Other: Self-assessment of dyspareunia
- Control (Waitlist) (Other): Participants will not have a PLR during the study period. They will be placed on a waitlist to receive the PLR at the end of the study period.
  Interventions: Other: Self-assessment of dyspareunia

INTERVENTIONS:
Device: Phallus Length Reducer — Phallus Length Reducer
  Other Names: OhNut
  Arms: Experimental (PLR)
Other: Self-assessment of dyspareunia — Use of a vaginal insert to self assess dyspareunia

SUMMARY:
The purpose of this study is to evaluate the acceptability and effectiveness of two tools that may help address the management of deep dyspareunia: 1) A phallus length reducer (PLR, brand name: Ohnut), consisting of 4 interconnected silicone rings worn externally over the penetrating object to reduce pain with deep penetration by allowing adjustable limitation of penetration depth, and 2) A vaginal insert for at home self-assessment of the extent and severity of deep dyspareunia.

DETAILED DESCRIPTION:
Background: Endometriosis is a gynecological condition characterized by the abnormal growth of endometrial like tissue outside of the uterus. The condition affects approximately 10% of reproductive-age females and can cause various types of pain, including chronic pelvic pain and deep dyspareunia (pelvic pain with deep sexual intercourse). Research has shown that individuals with endometriosis and dyspareunia have significantly reduced sexual quality of life, lower self-esteem, and impaired sexual function. Qualitative research has also demonstrated that many individuals with dyspareunia feel guilty about their pain, and often continue to engage in intercourse even when the pain is severe.

Aims and Hypotheses:

1. To measure the reduction in deep dyspareunia observed among people using the PLR with their partner. The investigators hypothesize that the PLR will be associated with a reduction in self-reported deep dyspareunia scores among participants randomized to the PLR intervention, compared to participants randomized to the waitlist control group. The measured reduction in deep dyspareunia will be used to power a future definitive trial.
2. To assess the acceptability of the phallus length reducer (PLR) for participants with endometriosis and their partners. The investigators hypothesize that both partners will indicate the PLR is acceptable on the self-reported questionnaire.
3. To explore whether an at-home assessment of dyspareunia is an acceptable and valid alternative to clinical measures. The investigators hypothesize that the at-home assessments of dyspareunia will be acceptable to participants and will yield results that are highly correlated with questionnaire-based and clinical assessments of this pain.

ELIGIBILITY:
Inclusion Criteria:

Patient

* 19 to 49 years of age
* Monogamous sexual partnership
* Sexually active or not sexually active due to deep dyspareunia
* Self-reported deep dyspareunia score ≥ 4/10
* Sexual partner who is willing to participate
* Willing to engage in penetrative sex at least once during the duration of the study

Partner

* 19 years of age or older
* Sexually active with a patient participant who has consented to participate in this study

Exclusion Criteria:

Patient

* Superficial dyspareunia score ≥ 4/10 (This is a potentially confounding variable; the PLR is not expected to affect introital pain)
* Current use of a PLR
* Inability to complete English-language questionnaires
* GAD-7 score ≥ 15
* PHQ-9 score ≥ 15
* Intense fear/anxiety in anticipation of, during, or as a result of vaginal intercourse

Partner

* Current use of a PLR
* Inability to complete English-language questionnaires

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants with endometriosis by definition are of the female sex but may self-identify with any gender identity. We are also recruiting their sexual partners, who may be of either sex, any gender identity.
Enrollment: 30 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of the phallus length reducer (PLR) | After 6 weeks of using the PLR
  Acceptability of the PLR as measured via questionnaire using a 5 point likert scale (1 = most negative/ worst/ strongly disagree, 5 = most positive/ best/ strongly agree)

SECONDARY OUTCOMES:
Severity of dyspareunia | Measured at baseline, before and after 6 weeks of using the PLR
  Self reported on an 11-point numeric rating scale (0 being no pain, 10 being worst pain imaginable)
Change in sexual function | Measured at baseline, before and after 6 weeks of using the PLR
  Change in sexual function as measured by Female Sexual Function Index (FSFI). This a brief, self-administered questionnaire to assess key dimensions of sexual function in women. The scale consists of 19 items that assess sexual function over the past four weeks and are scored from 1 to 5 (with 1 being the lowest report of desire and 5 being the highest).
Change in sexual distress | Measured at baseline, before and after 6 weeks of using the PLR
  Change in sexual distress as measured in Female Sexual Distress Scale-Revised (FSDS-R) This is a self-administered measure of female personal distress associated with sexual dysfunction. There are 13 questions. The range for each question is 0 (Never) to 4 (Always).
Change in level of general anxiety (GAD-7) | Measured at baseline, before and after 6 weeks of using the PLR
  Change in level of general anxiety as measured using the General Anxiety Disorder - 7 questionnaire. There are 7 questions. The range for each question is 0 (not at all) to 4 (nearly every day).
Change in level of general depression (PHQ-9) | Measured at baseline, before and after 6 weeks of using the PLR
  Change in level of general depression as measured using the Patient Health Questionnaire- 9 questionnaire. There are 9 questions. The range for each question is 0 (not at all) to 4 (nearly every day).
Acceptability of self-measurement of dyspareunia | After patient self-measurement of dyspareunia is complete (2 times during study)
  Acceptability of self-measurement of dyspareunia will be measured via questionnaire using 5 point likert scale (1 = most negative/ worst/ strongly disagree, 5 = most positive/ best/ strongly agree)
Validity of self-measurement of dyspareunia | Assessment and questionnaire administered 2 times, each one week apart, during the first 4 weeks of the study (to be assessed at week 2 and 3 of participant's menstrual cycle, which may vary)
  Dyspareunia score from the self-measurement will be compared to records of dyspareunia scores from physician performed pelvic exams. (11 point scale, 0 being no pain, 10 being worst pain imaginable)
Feasibility - Recruitment | Up to 6 months
  The proportion of potentially eligible individuals who were successfully contacted by the study team (response rate); the proportion of contacted individuals who were ineligible, declined to participate, and consented; the number of couples enrolled per month of active recruitment (recruitment rate).
Feasibility - Retention | Up to 6 months
  The proportion of enrolled participants who completed the study (retention rate).
Feasibility - Intervention Fidelity | Up to 6 months
  To evaluate protocol adherence we documented: the proportion of sexual encounters using the Ohnut per couple in the intervention group during the intervention period (intervention fidelity) and the proportion of missing data.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wahl K, Orr NL, Parmar G, Zhang SXJ, MacLeod RGK, Noga H, Albert A, Flannigan R, Brotto LA, Yong PJ. Ohnut vs waitlist control for the self-management of endometriosis-associated deep dyspareunia: a pilot randomized controlled trial. Sex Med. 2024 Aug 31;12(4):qfae049. doi: 10.1093/sexmed/qfae049. eCollection 2024 Aug. PMID 39220343
- [Derived] Zhang SXJ, MacLeod RGK, Parmar G, Orr NL, Wahl KJ, Noga H, Albert A, Flannigan R, Brotto LA, Yong PJ. Ohnut Versus a Waitlist Control for the Self-management of Endometriosis-Associated Deep Dyspareunia: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 27;12:e39834. doi: 10.2196/39834. PMID 36972117